CLINICAL TRIAL: NCT07085455
Title: The Effect of the Timing of Supplemental Parenteral Nutrition on the Prognosis of Critically Ill Patients (T-SPN): A Multicenter Randomized Controlled Trial
Brief Title: The Effect of the Timing of Supplemental Parenteral Nutrition on the Prognosis of Critically Ill Patients (T-SPN)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dong Zhang (Other)
Responsible Party: Sponsor-Investigator, Dong Zhang, chief physician, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T-SPN
Record Dates: First submitted 2025-07-07; First posted 2025-07-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Organ Dysfunction; Enteral Nutrition Intolerance; Inadequate Nutritional Intake
Keywords: Nutritional support; Supplementary parenteral nutrition; Early enteral nutrition; Severe patients; critical care; intensive care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to either the early supplemental parenteral nutrition (SPN) group or the late SPN group. Each group receives only one intervention throughout the study period, and outcomes are compared in a parallel manner.
Who Masked: Participant
Masking Description: Participants are blinded to group assignment to reduce expectation bias. The clinical staff administering the nutrition intervention are not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early SPN Group (Experimental): Patients in this group will receive supplemental parenteral nutrition (SPN) starting on day 4 after ICU admission, in addition to standard enteral nutrition (EN).
  Interventions: Dietary Supplement: Early Supplemental Parenteral Nutrition (SPN)
- Late SPN Group (Active Comparator): Patients in this group will receive SPN starting on day 8 after ICU admission, in addition to standard EN.
  Interventions: Dietary Supplement: Late Supplemental Parenteral Nutrition (SPN)

INTERVENTIONS:
Dietary Supplement: Early Supplemental Parenteral Nutrition (SPN) — SPN is initiated on ICU day 4 if enteral nutrition remains <50% of the target caloric requirement. Nutrition support is guided by protocol
  Arms: Early SPN Group
Dietary Supplement: Late Supplemental Parenteral Nutrition (SPN) — SPN is initiated on ICU day 8 if enteral nutrition remains <50% of the target caloric requirement. Nutrition support is guided by the same protocol as in the early SPN group.
  Arms: Late SPN Group

SUMMARY:
This multicenter, randomized controlled trial aims to evaluate whether early initiation of supplemental parenteral nutrition (SPN) (on day 4 of ICU admission) compared to late initiation (on day 8) can reduce 28-day all-cause mortality in critically ill patients. Secondary objectives include assessing the effects of early SPN on long-term functional outcomes (2-year EQ-5D-5L scores), mortality at various timepoints (ICU, 28-day, 90-day, 180-day, and 2-year), ICU length of stay, serum prealbumin levels (days 8 and 28), skeletal muscle measurements (diaphragm thickness, biceps, quadriceps, and rectus femoris cross-sectional area), incidence of ICU-acquired infections, adverse events (e.g., hyperglycemia, hypoglycemia, dyslipidemia, liver dysfunction), and ventilator-free days within 28 days.

Eligible patients are adults (≥18 years) with at least one organ failure (SOFA score ≥2) within 24 hours of ICU admission, expected to remain in the ICU for >72 hours, and unable to reach 50% of caloric target via enteral nutrition (EN) within the first 72 hours. A total of 946 patients will be enrolled and randomized to receive either early SPN (day 4) or late SPN (day 8) in addition to standard EN. Follow-up will include in-hospital assessments and telephone follow-ups at 28, 90, 180 days, and 2 years. The study hypothesizes that early SPN may improve short-term survival and nutritional/muscle status, though its impact on long-term quality of life remains to be determined.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled clinical trial designed to evaluate the impact of early supplemental parenteral nutrition (SPN) versus late SPN initiation on clinical outcomes in critically ill patients. The primary objective is to determine whether initiating SPN on day 4 of ICU admission, compared to day 8, can reduce 28-day all-cause mortality. Secondary objectives include assessing the effects of early SPN on functional status (2-year EQ-5D-5L), mortality at various time points (ICU, 28-day, 90-day, 180-day, and 2-year), ICU length of stay, nutritional markers (prealbumin levels on days 8 and 28), muscle mass indicators (diaphragm thickness, biceps, quadriceps, and rectus femoris cross-sectional area), incidence of ICU-acquired infections, ventilator-free days, and metabolic adverse events (such as hyperglycemia, hypoglycemia, hyperlipidemia, and liver dysfunction).

Baseline and clinical process data will be collected for all enrolled patients within the first 24 hours of ICU admission. This includes demographic data (age, sex, height, weight), severity scores (APACHE II, SOFA), and nutritional status.

Additional ICU-related data will be recorded, including:

Use of sedation and analgesia (yes/no), and Richmond Agitation-Sedation Scale (RASS) scores Use of vasopressors (yes/no), type of agent(s), dosage, and duration Vital signs, fluid balance, and mechanical ventilation status Contact information for patient surrogates or family members will be obtained to facilitate follow-up at Day 28, Day 90, Day 180, and 2 years after ICU admission.

Randomization Method A free recruitment model was adopted nationwide. The randomization plan was developed by the study statistician. Dynamic block randomization stratified by participating centers was used to allocate participants to either the early or late SPN group in a 1:1 ratio. The size of the permutation blocks was variable and blinded to the treating clinicians and nursing staff.

Statistical Analysis Continuous variables will be presented as mean ± standard deviation or median (interquartile range [IQR]) depending on distribution characteristics and compared using the independent samples t-test or Wilcoxon rank-sum test. Categorical variables will be reported as counts (percentages) and compared using Pearson's chi-square test or Fisher's exact test as appropriate. The Kaplan-Meier method and log-rank test will be used to compare 2-year survival between groups.

To assess whether baseline nutritional risk modifies the effect of the intervention, interaction terms will be incorporated into multivariate logistic regression models (for mortality) and linear regression models (for physical function). The significance of interaction terms will be tested using the likelihood ratio test.

Sensitivity analyses will treat NRS-2002 and mNUTRIC scores as ordinal variables and age as a continuous variable, repeating the regression models. Additionally, the Random Forest (RF) algorithm will be applied to explore potential nonlinear interactions between nutritional risk and intervention effects.

All statistical analyses will be conducted using JMP software (SAS Institute Inc., Cary, NC, USA). A two-sided P-value < 0.05 will be considered statistically significant, while the threshold for interaction terms will be set at P < 0.1 to enhance detection sensitivity.

Sample Size Calculation Sample size estimation was performed using PASS software. Based on previous literature, the 28-day mortality rate was assumed to be 8% in the early SPN group and 14% in the late SPN group. Assuming a 1:1 allocation ratio, a two-sided α of 0.05, and a statistical power (1-β) of 0.90, 430 patients were required per group. Accounting for a 10% dropout rate, the final total sample size was set at 946 patients.

ELIGIBILITY:
Inclusion Criteria：

1. Age ≥ 18 years
2. Failure of one or more organ systems within 24 hours of ICU admission, defined as Sequential Organ Failure Assessment (SOFA) score ≥ 2 in any single organ system
3. Expected ICU stay > 72 hours
4. Able to initiate early enteral nutrition (EN) within 48 hours of ICU admission
5. Enteral nutrition providing <50% of target caloric requirements within 72 hour Exclusion Criteria

1.Full oral intake or tolerance of full-dose EN; no need for SPN 2.Receiving palliative care or expected to die within 72 hours 3.Pregnant or lactating women 4.Long-term use of systemic corticosteroids or other immunosuppressive agents 5.Known malignancy currently receiving radiotherapy or chemotherapy 6.Contraindications to parenteral nutrition (PN) 7.Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2029-07-20 (Estimated)

PRIMARY OUTCOMES:
28-Day All-Cause Mortality | 28 days after ICU admission
  Death from any cause occurring within 28 days of ICU admission. This is a binary outcome (alive or dead). Lower mortality indicates better outcome.

SECONDARY OUTCOMES:
physical function score： EuroQol 5-Dimension 5-Level Questionnaire（EQ5D5L） | 28 days after ICU admission，90 days after ICU admission，180 days after ICU admission，2 years after ICU admission
  The EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) is a standardized instrument for measuring health-related quality of life. It includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels, and a visual analog scale (EQ-VAS) ranging from 0 to 100. The utility index score, calculated using the country-specific value set (e.g., China), typically ranges from <0 (worse than death) to 1 (perfect health). Higher scores indicate better health status.
ICU Length of Stay | Duration of ICU stay, from admission to discharge from ICU up to 28 days
  The number of days the patient remains in the intensive care unit (ICU), counted from the date of ICU admission to the date of ICU discharge. A higher number indicates longer ICU stay.
Serum Prealbumin Levels on Day 8, Day 28, Day 90, Day 180, and 2 Years | ICU day 8, day 28, and at 90 days, 180 days, and 2 years after ICU admission
  Serum prealbumin (transthyretin) concentrations will be measured at five time points (ICU day 8, day 28, and at 90 days, 180 days, and 2 years post-ICU admission). Venous blood samples will be used for laboratory analysis. Results will be reported in mg/dL. Higher levels indicate better nutritional status and recovery.
Muscle Ultrasound Measurements on Day 8, Day 28, Day 90, Day 180, and 2 Years | ICU day 8, day 28, and at 90 days, 180 days, and 2 years after ICU admission
  Muscle mass will be assessed by bedside ultrasound at five time points: ICU day 8, day 28, and at 90 days, 180 days, and 2 years post-ICU admission. Parameters include diaphragm thickness, biceps thickness, quadriceps thickness, and rectus femoris cross-sectional area. Ultrasound measurements will follow standardized anatomical landmarks and positioning. Higher values reflect greater muscle mass and better nutritional status.
Incidence of New Infections in the ICU | From ICU admission to ICU discharge up to 28 days
  The number of patients who develop new infections during their ICU stay. Only infections acquired after ICU admission will be counted. Definitions follow CDC/NHSN surveillance criteria, including ventilator-associated pneumonia (VAP), catheter-related bloodstream infection (CRBSI), urinary tract infection (UTI), etc. This is a binary outcome (infection: yes/no) or count variable (number of new infections).
Ventilator-Free Days Within 28 Days After ICU Admission | 28 days after ICU admission
  The number of days within the first 28 days after ICU admission during which the patient is alive and free from invasive mechanical ventilation. If the patient dies within 28 days, the ventilator-free days will be counted as 0. Higher values indicate better outcomes.
All-Cause Mortality at Multiple Time Points (ICU, 28days，90 days, 180 days, 2 years) | From ICU admission to 2 years after ICU admission
  All-cause mortality will be assessed at the following time points: during ICU stay, at 28 days, at 90 days, at 180 days, and at 2 years after ICU admission. Mortality status will be determined via hospital records or telephone follow-up. Lower mortality at each time point indicates better outcome.
The number of participants with Laboratory Safety Parameters and Liver Dysfunction | From ICU admission to Day 28
  Laboratory parameters including blood glucose, blood lipids (total cholesterol, triglycerides), serum creatinine, blood urea nitrogen, and transaminases (ALT, AST) will be measured during ICU stay and up to day 28. Liver failure will be diagnosed based on clinical and laboratory criteria (e.g., jaundice, coagulopathy, elevated transaminases and bilirubin). These indicators are used to assess metabolic tolerance and organ function related to nutrition interventions.

OTHER OUTCOMES:
Gastrointestinal Tolerance and Intestinal Function Indicators | Day 8 and Day 28 after ICU admission
  Gastrointestinal symptoms (including vomiting, abdominal distension, diarrhea, and gastric retention) will be recorded daily. Nutritional status will be assessed using a standardized nutritional scoring tool (e.g., NRS-2002 or mNUTRIC). Intestinal dysfunction will be graded according to validated ICU scoring criteria (e.g., ESICM WGAP guidelines and GIDS socre). These indicators reflect enteral tolerance and gut function during nutrition therapy.

CONTACTS AND LOCATIONS:
Overall Officials: dong zhang, Study Director — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No